CLINICAL TRIAL: NCT04002713
Title: Comparison of the Outcome of Choosing Free Anterolateral Thigh or Free Posterolateral Thigh Flap for Reconstruction in Patients With Head and Neck Cancer
Brief Title: Comparison of Choosing Free ALT or Free PMT for Reconstruction With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201900308B0
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Reconstructive Surgery; Head and Neck Cancer
Keywords: Anterolateral thigh (ALT); anteromedial thigh (AMT); free flap reconstruction; microsurgery; head and neck cancer; outcomes
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALT&AMT free flap reconstruction: Patients who underwent ALT or AMT free flap reconstruction after head and neck cancer surgery between March 1, 2008 and February 28, 2017
  Interventions: Other: ALT flap reconstruction; Other: AMT flap reconstruction

INTERVENTIONS:
Other: ALT flap reconstruction — Patients who underwent ALT free flap reconstruction after head and neck cancer surgery.
Other: AMT flap reconstruction — Patients who underwent AMT free flap reconstruction after head and neck cancer surgery.

SUMMARY:
This study was designed to compare the outcome of the anteromedial thigh (AMT) and anterolateral thigh (ALT) flaps in head and neck cancer reconstruction.

DETAILED DESCRIPTION:
To compare the results of the AMT and ALT flaps, this study aimed to compare their outcomes in head and neck cancer reconstruction under the condition of attenuating baseline patient and operative characteristics with the selection of propensity score-matched patient cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent ALT or AMT free flap reconstruction after head and neck cancer surgery between March 1, 2008 and February 28, 2017.

Exclusion Criteria:

* Patients whose data were missing will be excluded.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective study was performed on adult trauma patients from the registered free flap database and electric medical records of Kaohsiung Chang Gung Memorial Hospital, a 2,686-bed medical center in Southern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 1590 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
survival or failure | up to 6 months
  The primary free flap outcome was determined as its survival or failure.

SECONDARY OUTCOMES:
Complications | up to 6 months
  The second outcome was the associated complications (fistula, hematoma, partial necrosis, and wound infection).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan